CLINICAL TRIAL: NCT00839865
Title: Phase 1 Study of Herb Yuyang Ointment That Expressed Good Effect in Diabetic Foot Ulcer
Brief Title: Trial of Herb Yuyang Ointment to Diabetic Foot Ulcer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guiyang No.1 People's Hospital (Other)
Collaborators: Beijing University of Chinese Medicine (Other); Third Military Medical University (Other)
Responsible Party: Endocrinology Unit, Guiyang No.1 People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFL-2008-11; ISRCTN20081114; NCI-197-4128D; R01-020225-1
Expanded Access: Available
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Evidence-based evaluation; Multi-center randomized controlled clinical trials; Traditional Chinese Medicine; therapy; diabetic foot ulcer; clinical trails
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- herb ointment dressing change group (Experimental): This group of patients in the ointment dressing every 2 days until Wound Healing or 6 months
  Interventions: Drug: herb ointment
- Conventional dressing change group (No Intervention): This group of patients in the Conventional dressing every 2 days until Wound Healing or 6 months

INTERVENTIONS:
Drug: herb ointment — a kind of ointment made from herb
  Other Names: TANGZUYUYANGGAO
  Arms: herb ointment dressing change group

SUMMARY:
The purpose of this study is to determine if dressing change with a kind of herb Yuyang ointment is clinically more efficacious and safer than Conventional treatment in the treatment of diabetic foot ulcers.

DETAILED DESCRIPTION:
1. Developing a Document Retrieval strategy for clinical trials of Chinese medicine treatment of diabetic foot ulcer according to the research program(finished)
2. Selecting and Evaluating the above trials,developing a methodological quality evaluation criteria(finished)
3. extract information, verification, meta-analysis, sensitivity analysis and sub-group analysis(finished)
4. comprehensive evaluating the pros and cons evidences of traditional Chinese medicine, acupuncture and Chinese and Western combined medicine with the treatment of diabetic foot of (finished)
5. we find dress change with a certain kind of herb ointment is very effective and safe to diabetic foot ulcers.The following step is randomized controlled multicenter clinical trial to verify it's efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

* In-patient or out-patient patients diagnosed with diabetic foot ulcers
* Gangrene or ulceration occurred more than 3 weeks
* Over 18 years of age
* Gender-open
* The type of diabetes (type 1 or type 2) open
* Patients receive a written informed consent to participate in the trial

Exclusion Criteria:

* Serious complications of heart, liver, lung, kidney damage
* Malignant tumors
* Allergy for Chinese medicine used
* Pregnant women and breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to determine the effect of this ointment on the incidence of complete wound closure. | 6 months

SECONDARY OUTCOMES:
Secondary objectives include: evaluating the acceleration of ulcer closure or facilitation of surgical closure, reduction of ulcer surface area over time, reduction in complications, the quality of life and it's safety. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Shufa, doctor, Study Chair
Locations (1):
- endocrinology unit,No.1 people's hospital of Guiyang City, Guiyang, Guizhou, China

REFERENCES:
- [Background] Leung PC, Wong MW, Wong WC. Limb salvage in extensive diabetic foot ulceration: an extended study using a herbal supplement. Hong Kong Med J. 2008 Feb;14(1):29-33. PMID 18239240